CLINICAL TRIAL: NCT05623852
Title: A Phase II Trial for Oligo-Fucoidan in Cancer Cachexia and Sarcopenia
Brief Title: The Impact of Oligo-Fucoidan in Cancer Cachexia and Sarcopenia
Acronym: OFCS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Collaborators: Asia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB109-195-A
Record Dates: First submitted 2022-04-07; First posted 2022-11-21 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-04

CONDITIONS: Cachexia
Keywords: Cachexia; sarcopenia; fucidan
MeSH Terms: conditions — Cachexia; Sarcopenia | interventions — fucoidan

STUDY DESIGN:
Intervention Model Description: Study Type : Interventional (Clinical Trial) Actual Enrollment : 100 participants Allocation: Randomized Intervention Model: Parallel Assignment, matching sex, age, and performance status
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Fucoidan arm (Experimental): It is recommended to consume on an empty stomach, 2 servings per day, a total of 8 tablets, which can be eaten at one time or in divided doses. If it is difficult to swallow, the powder in the capsule can also be taken out and mixed with food or liquid food.
  Interventions: Dietary Supplement: fucoidan
- Arm B, Observational arm (No Intervention): observation

INTERVENTIONS:
Dietary Supplement: fucoidan — It is recommended to consume on an empty stomach, 2 servings per day, a total of 8 tablets, which can be eaten at one time or in divided doses. If it is difficult to swallow, the powder in the capsule can also be taken out and mixed with food or liquid food.
  Arms: Arm A: Fucoidan arm

SUMMARY:
Fucoidan also ameliorates tumour and chemotherapy-induced muscle atrophy and -related cachectic symptoms in vivo and in vitro. To evaluate the effect of fucoidan in cancer cachexia or sarcopenia in cancer patients.

DETAILED DESCRIPTION:
Cancer cachexia is characterized by anorexia, skeletal muscle atrophy, and systemic inflammation. Fucoidan extracted from brown algae exhibits anti-inflammatory and anticancer activities. In addition, fucoidan also ameliorates tumour and chemotherapy-induced muscle atrophy and -related cachectic symptoms in vivo and in vitro. To evaluate the effect of fucoidan in cancer cachexia or sarcopenia in cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed patients with stage III-IV non-small cell lung cancer, colorectal carcinoma, head and neck cancer, nasopharyngeal cancer, or pancreatic carcinoma, who are not eligible for surgery, and interventional treatment .
2. Chemotherapy regimen include platinum-based drugs and Gemcitabine based drugs;
3. For patients who are being treated with chemotherapy, the chemotherapy regimen should be confined to the regimens specified in the protocol; and the chemotherapy regimen, in general, are not allowed to be changed during the study period;
4. Patients are conscious and able to cooperate with the doctor to complete the disease-related examinations and evaluations;
5. ECOG performance status (PS) 0-3 for those who are not treated with chemotherapy; and ECOG PS 0-2 for those who are being treated with chemotherapy;
6. Expected survival period is more than 3 months;
7. Male or female aged 20 - 90 years;
8. Patients who are willing to participate in the study and sign the informed consent form.

Exclusion Criteria:

1. Patients who are being treated with chemotherapy, the chemotherapy regimen is not among the regimens specified in the protocol;
2. Patients with cachexia caused by other reasons, e.g. severe hepatic dysfunction [Aspartate transaminase(AST)/Cerealthirdtransaminase(ALT) >5 times the ULN], severe renal dysfunction (Cr >1.5 times the ULN), uncontrolled thyroid disease, New York Heart Association (NYHA) class III-IV heart failure, AIDS etc.;
3. Any condition that may hinder the subject's completion of the study, including but not limited to severe uncontrollable organic diseases or infection, unstable angina pectoris, congestive heart failure, etc.;
4. Known or suspected diagnosis of metastatic encephaloma;
5. Patients present with an ECOG score>2 and require treatment of chemotherapy;
6. Patients who are currently included in other clinical trials on antineoplastic drugs;
7. Patients who are not able to provide the Informed Consent Form (ICF);
8. Expected survival period is less than 4 months;
9. Female patient is pregnant or breast-feeding, and those patients at childbearing age who are not willing to use methods of contraception (including males);
10. Patients with symptomatic, uncontrolled nervous disorders, mental illness or psychiatric disorder;
11. Any condition, in the investigator's opinion, is not in the best interest of the subject (e.g., harming the subject's health) or potentially interferes with the evaluation of treatment according to this protocol.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-01-30 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Body Weight | 0 day, 60th day, and 90th day Body weight change
  Body Weight Change. (kilograms)

SECONDARY OUTCOMES:
Lean Mass Measured by Densitometry | 0 day, 60th day, and 90th day
  Lean body mass measured by DEXA. Percentage of change day 90, 60-baseline. (%)
Muscle Strength as Measured by Grip Strength. | 0 day, 60th day, and 90th day
  Dominant hand grip strength day 90, 60 - percent change from baseline (%)
Quality of life as assessed using the FACIT-F Patient Reported Outcome assessments | 0 day, 60th day, and 90th day
  Quality of life as assessed using the FACIT-F Patient Reported Outcome assessments - percentage of change day 90, 60-baseline (with a range from 0 to 52)
Appetite | 0 day, 60th day, and 90th day
  Appetite measured by a visual analogue scale ASAS. Percentage of change day 90, 60-baseline (providing a range of scores from 0-100)
Resting Energy Expenditure | 0 day, 60th day, and 90th day
  % change between day 90, 60 and baseline (%)
Functional Performance | 0 day, 60th day, and 90th day
  Functional performance using stair-climbing power day 90, 60 percent change from baseline (continuous variable ) Power = Work/time Power = (acceleration due to gravity) x mass x distance/time
1-repetition Max. Strength | 0 day, 60th day, and 90th day
  leg extension - percentage of change day 90, 60 to baseline (%)
Food Diary Calorie Count | 0 day, 60th day, and 90th day
  change between day 90, 60 and baseline (continuous variable, t-test)
Biomarkers TNF-alpha, IL-6, IGF-1 and IGFBP-3. | 0 day, 60th day, and 90th day
  change between day 90, 60 and baseline(continuous variable, t-test)

CONTACTS AND LOCATIONS:
Overall Officials: Szu-Yuan Wu, Principal Investigator — Asia University, Taiwan
Locations (2):
- Taiwan (2):
  - Asia University, Taichung, Please Select
  - Szu-Yuan Wu, Taipei, Please Select

IPD SHARING:
Plan to Share IPD: Yes
study completed
Supporting Information: Study Protocol
Time Frame: data will become available on April 30 2022.
Access Criteria: requirement with official application